CLINICAL TRIAL: NCT05299203
Title: Phase Ia/Ib Clinical Trial of Sapropterin Dihydrochloride Tablets in the Prevention and Treatment of Radiation-induced Skin Reactions in Intensity Modulated Radiotherapy for Head and Neck Squamous Cell Carcinoma (Including Nasopharyngeal Carcinoma)
Brief Title: BH4 in the Prevention and Treatment of Radiation-induced Skin Reactions for Head and Neck Squamous Cell Carcinoma (Including Nasopharyngeal Carcinoma)
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Xingchen Peng, PhD, Professor, West China Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ChiCTR2100054693
Record Dates: First submitted 2022-02-03; First posted 2022-03-28 (Actual); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Head and Neck Squamous Cell Carcinoma
Keywords: head and neck squamous cell carcinoma; nasopharyngeal carcinoma; radiation dermatitis; Sapropterin dihydrochloride; BH4
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Nasopharyngeal Carcinoma; Radiodermatitis | interventions — sapropterin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dose Escalation and Expansion (Experimental): In the dose escalation phase, 9 patients will be included in 3 groups with 3 patients as one group. In the dose expansion phase, the concentration of Sapropterin dihydrochloride tablets (BH4) aqueous solution will be performed according to the effective concentration of dose escalation phase, and 9 patients will be enrolled.
  Interventions: Drug: Sapropterin dihydrochloride tablets

INTERVENTIONS:
Drug: Sapropterin dihydrochloride tablets — dose escalation phase (BH4) aqueous solution is sprayed onto the skin of all radiotherapy areas, 3 times a day until two weeks after the end of radiotherapy.

SUMMARY:
Head and neck squamous cell carcinoma (include nasopharyngeal carcinoma) is one of the most common malignant tumor in China, and radiotherapy is the main treatment method. Radiation-induced dermatitis is one of the most common complications of head and neck squamous cell carcinoma patients during radiotherapy. Severe radiation dermatitis will cause secondary infection, severe pain, and even lead to the interruption of radiotherapy. On the one hand, it will affect the efficacy of tumor treatment, which may affect the long-term survival of patients, and on the other hand, it will also seriously affect the quality of life of patients. Tetrahydrobiopterin（BH4）, also known as sapropterin, has been shown not only to reduce the severity of acute radiation dermatitis but also to enhance the repair of skin injury in animal experiments. It may be a new approach and method for the prevention and treatment of radiation-induced dermatitis

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed diagnosis of head and neck squamous cell carcinoma (including nasopharyngeal carcinoma).
2. Age ≥ 18 years old, ≤ 80 years old.
3. Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
4. Head and neck radiotherapy alone or concurrent chemoradiotherapy, radiotherapy using intensity modulated radiotherapy.
5. Blood routine examination: hemoglobin ≥ 100g/L, platelet count ≥ 75×10^9/L, white blood cell count ≥ 3.0×10^9/L, absolute neutrophil count ≥ 1.5×10^9/L. Blood biochemistry: total bilirubin≤1.5 upper limit of normal (ULN), alanine aminotransferase (ALT) and aspartate aminotransferase (AST)≤2.5 ULN, serum creatinine ≤1.5 ULN or creatinine clearance rate >=60ml/min.
6. Have signed informed consent form.

Exclusion Criteria:

1. Allergic to the components of Sapropterin dihydrochloride tablets or severe allergic constitution.
2. Poor compliance.
3. Pregnant or breastfeeding.
4. Any previous radiotherapy to the head and neck region.
5. Patients deemed unsuitable for the study by the investigator (concomitant with any other serious disease)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2022-05 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Radiation dermatitis grading change from the baseline to the 4 weeks after radiotherapy | Assessment is performed two weeks before radiotherapy, once a week during radiotherapy, the day at the end of radiotherapy, once a week for 4 weeks after radiotherapy.
  Radiation dermatitis is assessed according to the CTCAE 5.0 radiation dermatitis grading scale

SECONDARY OUTCOMES:
Subjects' quality of life score change from the baseline to the 4 weeks after radiotherapy | Assessment is performed two weeks before radiotherapy, the day at the end of radiotherapy, 2 weeks after radiotherapy, 4 weeks after radiotherapy.
  Subjects' quality of life is assessed according to the Spitzer Quality-of-Life Index (SQLI)

CONTACTS AND LOCATIONS:
Overall Officials: Xingchen Peng, Ph.D, Principal Investigator — West China Hospital